CLINICAL TRIAL: NCT05679791
Title: Comparative Study of Static and Dynamic Hand Grip Endurance With Correlation of Deep Breathing Among Pregnant Women; A Cross-sectional Study
Brief Title: Comparative Study of Static and Dynamic Hand Grip Endurance in Pregnancy
Status: Completed | Type: Observational
Sponsor: Central Park Medical College (Other)
Collaborators: Shalamar Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, Mirza Zeeshan Sikandar, Principal Investigator, Central Park Medical College
Other Study IDs: SSAHS-IRB/AL/34/2022
Record Dates: First submitted 2023-01-03; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Hand Grasp; Pregnancy Related
MeSH Terms: interventions — Muscle Strength Dynamometer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Device: Dynamometer
- Group 2
  Interventions: Device: Dynamometer

INTERVENTIONS:
Device: Dynamometer — to assses hand grip

SUMMARY:
Background: Physiology of the mother, changes constantly during pregnancy including reduced HGS that is require for carrying the child after delivery. Activities of daily living require manual gripping tasks that require dynamic and static contractions. Predictor of upper extremity function is Hand Grip Strength and handgrip endurance. Screening of hand grip strength during antenatal care is still uncommon.

Objectives: To compare static and dynamic hand grip endurance in pregnant females and to find its correlation with deep breathing.

Material and Methods: The study recruited 40 participants of primi-gravida of 1st and 2nd trimester, between ages 20 and 35 years from SHALAMAR GYNAE OPD. The participants assigned to the groups (Group 1: with DB, Group 2: without DB) based on their trimester and gravidity. Static and dynamic endurance assessed using hand held dynamometer.

Key words: Pregnancy, deep breathing, trimester, endurance, peak grip endurance

ELIGIBILITY:
Inclusion Criteria:

* primigravida

Exclusion Criteria:

* multigravida
* Cardiac patients

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: Females
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
hand grip in pregnancy | feb 2022 to aug 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Central Park Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes